CLINICAL TRIAL: NCT03648125
Title: Influence of Dental Occlusion on the Performance of High Level Rowers (IODPR)
Acronym: IODPR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited time between the beginning and the end of the inclusions, only 7 high level rowers available within the time compatible with research realization
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC17_8823_IODPR
Record Dates: First submitted 2018-05-25; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Dental Occlusion, Traumatic
Keywords: young elite rowers
MeSH Terms: conditions — Dental Occlusion, Traumatic

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, randomized, open-label, cross-over study. Randomization applies on the order of the training sessions "with" or "without" occlusal disturbance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rowing training session (Other): Power tests, balance and tonicity tests are performed eyes opened and eyes closed :
  * with artificial occlusal disturbance and
  * without artificial occlusal disturbance
  Interventions: Device: with artificial occlusal disturbance; Device: without artificial occlusal disturbance

INTERVENTIONS:
Device: with artificial occlusal disturbance — A silicon artificial occlusal disturbance is made from a mould of the rowers mouth and placed in the mouth during the training session.
  With artificial occlusal disturbance : Maximal Intercuspal Occlusion (MIO) with silicone splint increases the vertical dimension of occlusion of 1, 2 and 4 mm.
Device: without artificial occlusal disturbance — The training session is performed without occlusal disturbance

SUMMARY:
Monocentric, prospective, randomized, open-label, cross-over study.

DETAILED DESCRIPTION:
Current literature data suggest that dental occlusion has an influence on postural control in the general population, and more markedly in high-level athletes. The link between dental occlusion and the postural stability of top athletes has been studied in several disciplines such as basketball, shooting, golf and running. There is currently no data in the field of rowing. But this sport requires optimal postural control for synchronous and symmetrical muscle solicitation.

The present study aims to evaluate the influence of dental occlusion on postural stability and the performance of high level rowers.

Our assumptions are as follows:

* Occlusal disturbance alters the muscular power developed by high level rowers
* occlusal disturbance alters the static postural stability of high level rowers

ELIGIBILITY:
Inclusion Criteria:

* High level rower, part of the Lille Rowing Hope Pole;
* At least 15 years old;
* Training at the Centre de Ressources, d'Expertise et de Performance Sportive (CREPS) de Wattignies during the period from 01/09/2017 to 31/10/2017;
* Having at least 28 natural or prosthetic teeth in occlusion;
* Not having consumed alcohol in the last 24 hours before the recordings;
* whose parents have given free, informed and written consent for minors;
* Having given free and informed consent, in writing supplemented by the consent of at least one holder of parental authority, if he is a minor;
* Affiliated, himself or through his parents if he is a minor, to a social security scheme.

Exclusion Criteria:

* Current antecedent(s) or pathology(s) likely to disturb the balance: neurological, ear nose and throat, ophthalmological, orthopedic;
* Temporomandibular joint disorder (s) (pain and / or noise);
* Orofacial symptoms (headache, tinnitus, facial myalgia, bruxism);
* Dental and / or periodontal care in progress;
* Chronic pain requiring daily use of analgesics for more than three months;
* Pregnant or lactating woman;
* Concurrent participation in another study;
* Major persons subject to legal protection (safeguard of justice, guardianship, tutorship) and persons deprived of their liberty.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Muscular power | At the time of inclusion
  Muscular power (in Watts) developed by the high level rowers with the "leg press" test on a "Dyno concept 2" machine, with and without artificial occlusal disturbance. Each test lasts 30 seconds. The sequence consists in 2 tests and is performed twice with a resting period of 1 min between each recording.

SECONDARY OUTCOMES:
Surface of the pressure center of the rower's feet | At the time of inclusion
  Each test lasts 51.2 seconds. The sequence consists in 10 tests and is performed twice with a resting period of 1 min between each recording.
  During each test, the projected sway area (in mm², the area of the confidence ellipse containing 90% of the sampled positions of the foot pressure center on the statokinesigram) is extracted from the stabilometric platform
Velocity of the pressure center of the rower's feet | At the time of inclusion
  Each test lasts 51.2 seconds. The sequence consists in 10 tests and is performed twice with a resting period of 1 min between each recording.
  During each test, the sway velocity (in mm/s) is calculated as the speed of displacement of the center of pressure of the foot as a function of the average position on the antero-posterior axis of the statokinesigram.
Tonicity of the para-vertebral muscles | At the time of inclusion
  Tonicity of the para-vertebral muscles is evaluated with the postural test of Posterior-superior iliac spines (PSIS) with and without artificial occlusal disturbance. This PSIS test is performed eyes opened, in MIO position with and without artificial occlusal disturbance,
  The sequence of two tests is performed twice. During this test, the endpoint is qualitative: operator asymmetric thumbs' ascension reflecting asymmetric contraction of paravertebral muscles (abnormal response) or not (normal response).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MD RAVALEC, Principal Investigator — Rennes University Hospital
Locations (1):
- CREPS de Wattignies, Wattignies, Hauts-de-France, France